CLINICAL TRIAL: NCT02769195
Title: Utility of a Measure of Lupus Low Disease Activity State (LLDAS) in SLE: Pooled Analysis of the HGS1006-C1056 (BLISS-76) and HGS1006-C1057 (BLISS-52) Trials
Brief Title: Utility of a Measure of Lupus Low Disease Activity State (LLDAS) in SLE
Status: Completed | Type: Observational
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Dr Emily Pei Xuan Ong, Dr, Monash University
Other Study IDs: CF16/684 - 2016000335; CSDR-1320 (Other: GSK)
Record Dates: First submitted 2016-04-12; First posted 2016-05-11 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a secondary, pooled analysis of two completed phase 3 clinical trials:

(i) GSK-HGS1006-C1056 (BLISS-76): A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, 76-Week Study to Evaluate the Efficacy and Safety of Belimumab (HGS1006, LymphoStat-B™), a Fully Human Monoclonal Anti-BLyS Antibody, in Subjects with Systemic Lupus Erythematosus (SLE); and,

(ii) GSK-HGS1006-C1057 (BLISS-52): A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, 52-Wk Study to Evaluate the Efficacy and Safety of Belimumab (HGS1006, LymphoStat-B™), a Fully Human Monoclonal Anti-BLyS Antibody, in Subjects With Systemic Lupus Erythematosus (SLE)

The study will assess the discriminant validity of a proposed measure of low disease activity (the Lupus Low Disease Activity State, LLDAS) in patients with SLE.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a multisystem autoimmune disease with an estimated incidence of 5-50 cases per 100,000 people. Despite advances in therapy, there is still significant mortality and morbidity associated with this disease. There have been no clearly defined treatment goals in SLE, hindering the development of treat to target approaches and evaluation of new therapies. Although remission is aimed for, it rarely occurs. A more achievable clinical state and treatment goal of low disease activity has been described recently and a preliminary single centre validation study has demonstrated its association with improved outcomes. This endpoint is termed Lupus Low Disease Activity State (LLDAS).

The proposed study will assess the discriminant validity of the proposed LLDAS criteria in a clinical trial dataset. The objective of the research is to validate the Lupus Low Disease Activity State (LLDAS) tool as a study endpoint in SLE. The data available from the belimumab BLISS trials will be used to evaluate the LLDAS score.

The outcome of these studies will be validation of the LLDAS instrument in a clinical trial dataset, for the first time. This will allow future studies to consider incorporating LLDAS attainment as a trial endpoint, for example allowing comparison of frequency of achieving LLDAS to discriminate between treatments.

The findings will be interpreted using statistical methods and will be published / presented to the public and to peers via peer-reviewed publications, conference presentations, and where relevant the lay media.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of SLE by ACR criteria.
* Active SLE disease.
* Autoantibody-positive.
* On stable SLE treatment regimen.

Key Exclusion Criteria:

* Pregnant or nursing
* Have received treatment with any B cell targeted therapy.
* Have received treatment with a biological investigational agent in the past year.
* Have received IV cyclophosphamide within 180 days of Day 0.
* Have severe lupus kidney disease.
* Have active central nervous system (CNS) lupus.
* Have required management of acute or chronic infections within the past 60 days.
* Have current drug or alcohol abuse or dependence.
* Have a historically positive test or test positive at screening for HIV, hepatitis B, or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of the BLISS-76 and BLISS-52 Phase 3 clinical trials. Refer to ClinicalTrials.gov records NCT00410384 and NCT00424476 for further information about these studies.
Sampling Method: Probability Sample
Enrollment: 1684 (Actual)
Dates: Start 2016-04; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who attain the Lupus Low Disease Activity State (LLDAS) | 52 weeks
  A composite end-point involving SLEDAI-2K ≤4 with no reported renal, central nervous system, cardiopulmonary, vasculitis or gastrointestinal activity and no reported fever, hemolytic anemia or new disease activity since last assessment), SELENA-SLEDAI Physician Global Assessment ≤1, a current prednisolone dose of ≤7.5 mg daily and tolerance of maintenance doses of immunosuppressive drugs and approved biologic agents.

SECONDARY OUTCOMES:
Number of patients achieving a SLE Responder Index (SRI) Response | 52 weeks
  a ≥ 4 point reduction from baseline in SELENA-SLEDAI score, and no worsening (increase of < 0.30 points from baseline) in PGA, and no new BILAG A organ domain score or 2 new BILAG B organ domain scores compared with baseline.
  SELENA SLEDAI is calculated from 24 individual descriptors; 0 indicates inactive disease and the maximum theoretical score is 105; scores > 20 are rare. PGA is a visual analog scale scored from 0 to 3 (1=mild, 2=moderate, 3=severe). BILAG uses a single score for each of the 8 organ domains; range is from severe to no disease (A to E).

IPD SHARING:
Plan to Share IPD: No
This study is a secondary analysis of two existing clinical trial datasets. Anyone who wants to use the data should contact the primary study sponsor (GSK) via their data sharing website: https://clinicalstudydatarequest.com/

REFERENCES:
- [Background] Franklyn K, Lau CS, Navarra SV, Louthrenoo W, Lateef A, Hamijoyo L, Wahono CS, Chen SL, Jin O, Morton S, Hoi A, Huq M, Nikpour M, Morand EF; Asia-Pacific Lupus Collaboration. Definition and initial validation of a Lupus Low Disease Activity State (LLDAS). Ann Rheum Dis. 2016 Sep;75(9):1615-21. doi: 10.1136/annrheumdis-2015-207726. Epub 2015 Oct 12. PMID 26458737
- [Background] Oon S, Huq M, Golder V, Ong PX, Morand EF, Nikpour M. Lupus Low Disease Activity State (LLDAS) discriminates responders in the BLISS-52 and BLISS-76 phase III trials of belimumab in systemic lupus erythematosus. Ann Rheum Dis. 2019 May;78(5):629-633. doi: 10.1136/annrheumdis-2018-214427. Epub 2019 Jan 24. PMID 30679152